CLINICAL TRIAL: NCT04780256
Title: Retrospective Study of Efficacy and Safety of the Endoscopic Removal of Cancerous and Precancerous Lesions of the Upper and Lower Digestive Tract
Brief Title: Endoscopic Resection of Gastrointestinal Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: CORE 3
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-01

CONDITIONS: Endoscopic Mucosal Resection; Endoscopic Submucosal Dissection; Gastric Neoplasm; Colonic Neoplasms; Esophageal Neoplasms; Duodenal Neoplasms
Keywords: Endoscopic mucosal resection (EMR); Endoscopic submucosal dissection (ESD); Endoscopic full thickness resection (EFTR); Colorectal ESD; Colorectal EMR
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Duodenal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Endoscopic resection — The endoscopic resection is the procedure that allows to remove cancerous or precancerous conditions of digestive tract. Endoscopic resection can be preformed by several techniques:
  1. Endoscopic mucosal resection (EMR): it allows to remove mucosal lesions
  2. Endoscopic submucosal dissection: it allows to remove mucosal lesions that involved submucosal layer and large lesions
  3. Full-thickness resection: it allows to remove infiltrating lesions by the resection of a little piece of the entire gastrointestinal wall

SUMMARY:
The study aims to retrospectively investigate the endoscopic resection procedures of cancerous and precancerous lesions of the upper and lower digestive tract in order to evaluate the efficacy and safety outcomes and to compare different resection techniques. In particular, the resection techniques investigated will be mucosectomy, en bloc and piecemeal, endoscopic submucosal dissection (ESD) and its variants, full-thickness resection. The anatomical districts involved will be the esophagus, stomach, duodenum, colon and rectum.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* all patients who have undergone endoscopic resection of an upper or lower digestive tract tumor

Exclusion Criteria:

* age under 18
* inability to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients> 18 years of age who have undergone endoscopic resection of cancerous or pre-cancerous lesions of the digestive tract will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
en bloc resection rate | one month
  the en bloc resection is the ability to remove the neoplasia in a single piece
complete resection rate | one month
  the complete resection is the ability to remove the neoplasia with clear margins (R0)
recurrence rate | one year
  recurrence is the recurrence of the neoplasm at the resection site during follow-up

SECONDARY OUTCOMES:
adverse events rate | one month
  complication rate, early or late, related to the procedure used for endoscopic resection
costs | one month
  evaluation of the costs incurred to perform the endoscopic resection

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS-AUSL Reggio Emilia, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cecinato P, Lisotti A, Azzolini F, Lucarini M, Bassi F, Fusaroli P, Sassatelli R. Left colonic localization, non-granular morphology, and pit pattern independently predict submucosal fibrosis of naive colorectal neoplasms before endoscopic submucosal dissection. Surg Endosc. 2023 Apr;37(4):3037-3045. doi: 10.1007/s00464-022-09828-0. Epub 2022 Dec 21. PMID 36542136